CLINICAL TRIAL: NCT05243940
Title: Recovery Parameters and Nociception Levels in Opioid-free Versus Opioid Based Anesthesia for Thyroidectomy
Brief Title: Opioid-free Anesthesia in Thyroidectomies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: annie-rammi
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Pain, Post Operative; Pain, Acute; Pain, Chronic; Pain, Neuropathic; Pain, Nociceptive; Ketamine; Dexmedetomidine; Lidocaine; Fentanyl; Analgesia; Analgesics; Analgesics Non-narcotic
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Chronic Pain; Neuralgia; Nociceptive Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine-ketamine-lidocaine (DKL) group (Active Comparator): combination of dexmedetomidine-ketamine-lidocaine in one syringe
  Interventions: Drug: dexmedetomidine-ketamine-lidocaine (DKL)
- remifentanil (control) group (Active Comparator): remifentanil infusion (TCI Minto protocol)
  Interventions: Drug: remifentanil infusion

INTERVENTIONS:
Drug: dexmedetomidine-ketamine-lidocaine (DKL) — patients will be administered 0.25 mcg/kg Dexmedetomidine in 100 mL of normal saline within 10 minutes. Followingly, they will receive 1 mL/10 kg of the solution containing ketamine, lidocaine and dexmedetomidine at predefined concentrations. As maintenance, they will be receiving
  1mL/10kg/h of the aforementioned solution.
  Arms: dexmedetomidine-ketamine-lidocaine (DKL) group
Drug: remifentanil infusion — remifentanil infusion under the Minto model (target controlled infusion-TCI aiming at 4ng/ml blood concentration
  Arms: remifentanil (control) group

SUMMARY:
The aim of this study will be to investigate the effect of an opioid-free anesthesia regimen with a mixture of dexmedetomidine-lidocaine-ketamine in the same syringe versus fentanyl analgesia in elective thyroidectomies. Recovery parameters and nociception levels throughout the operation will be evaluated

DETAILED DESCRIPTION:
In the usual anesthetic practice opioids are often administered in the perioperative period for intraoperative analgesia to control the nociceptive pathway of pain and post-surgical pain management. However, in recent years, opioid Free Anesthesia (OFA) has become increasingly popular, in which opioid administration is avoided intraoperatively and minimized or avoided in the postoperative period.

Opioid-free anesthesia (OFA) has been shown to decrease postoperative complications associated with opioids, include sedation, dizziness, nausea, vomiting, constipation, physical dependence, tolerance, and respiratory depression.

Therefore, the investigators aim to perform this study to determine a goal-directed approach, which targets adequate antinociception (e.g., by measuring nociceptive/antinociceptive balance) that could reduce the negative effects of excessive drug infusion, prevent postoperative pain and improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* American Society of Anesthesiologists (ASA) classification I-II
* elective thyroidectomy

Exclusion Criteria:

* body mass index (BMI) >35 kg/m2
* contraindications to local anesthetic administration
* systematic use of analgesic agents preoperatively
* chronic pain syndromes preoperatively
* neurological or psychiatric disease on treatment
* pregnancy
* severe hepatic or renal disease
* history of cardiovascular diseases/ arrhythmias/ conduction abnormalities
* bradycardia(<55 beats/minute)
* drug or alcohol abuse
* language or communication barriers lack of informed consent

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
change from baseline in Quality of Recovery (QoR)-40 score after surgery | 24 hours postoperatively
  The QoR-40 is used to measure functional recovery and has been validated in patients undergoing general surgical procedures. Five general quality-of-recovery dimensions are measured within the QoR-40: physical comfort (12 items), emotional state (9 items), physical independence (5 items), psychological support (7 items), and pain (7 items). Each item is graded on a five-point Likert scale, and the global scores range from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery)
pain score on arrival to Post-Anesthesia Care Unit (PACU) | immediately postoperatively
  pain score by the use of Numeric Rating Scale (NRS) on arrival to PACU, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score at discharge from Post-Anesthesia Care Unit (PACU) | at discharge from Post Anesthesia Care Unit (PACU), approximately 1 hour postoperatively
  pain score by the use of Numeric Rating Scale (NRS) at discharge from PACU, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 3 hours postoperatively | 3 hours postoperatively
  pain score by the use of Numeric Rating Scale (NRS) 3 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 6 hours postoperatively | 6 hours postoperatively
  pain score by the use of Numeric Rating Scale (NRS) 6 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 24 hours postoperatively | 24 hours postoperatively
  pain score by the use of Numeric Rating Scale (NRS) 24 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
Nociception Level | intraoperatively
  Nociception Level as measured via the NOL (Nociception Level) index, whose values vary from 0 to 100 (100 represents the maximum level of nociception and 0 represents total absence of nociception). The aim of the current study will be to record percentage of operative time during which NOL levels will be <25

SECONDARY OUTCOMES:
remifentanil requirement during anesthesia | intraoperatively
  rescue remifentanil required intraoperatively to maintain systolic arterial blood pressure and heart rate within the 20% of baseline value
Post Anesthesia Care Unit (PACU) duration of stay | immediately postoperatively
  duration of patient stay at PACU
sedation on arrival to Post-Anesthesia Care Unit | immediately postoperatively
  sedation will be assessed with a 5-point sedation scale, where: 1, patient perfectly conscious; 2, patient feels a little drowsy; 3, patient seems to be sleeping but immediately reacts to verbal stimulation; 4, patient seems to be sleeping but slowly reacts to verbal stimulation and 5, patient seems to be sleeping and does not react to verbal stimulation but does react to a stimulus such as shaking or pain
sedation at discharge from Post-Anesthesia Care (PACU) Unit | at discharge from Post Anesthesia Care Unit (PACU), approximately 1 hour postoperatively
  sedation will be assessed with a 5-point sedation scale, where: 1, patient perfectly conscious; 2, patient feels a little drowsy; 3, patient seems to be sleeping but immediately reacts to verbal stimulation; 4, patient seems to be sleeping but slowly reacts to verbal stimulation and 5, patient seems to be sleeping and does not react to verbal stimulation but does react to a stimulus such as shaking or pain
time to first request for analgesia | during stay in Post-Anesthesia Care Unit (PACU), approximately 1 hour postoperatively
  the time for the first patient request for analgesia will be noted
morphine consumption in Post-Anesthesia Care Unit (PACU | immediately postoperatively
  mg of morphine requested during patient PACU stay
tramadol consumption in the first 48 hours | 48 hours postoperatively
  patients will be followed for cumulative tramadol consumption for 48 hours postoperatively
sleep quality | 24 hours postoperatively
  subjective evaluation of sleep quality by patients, based on a sleep questionnaire (evaluation of sleep duration, number of nocturnal awakenings and marking of sleep quality)
first mobilization after surgery | 24 hours postoperatively
  patients will be questioned regarding the time at which they mobilized after surgery
satisfaction from postoperative analgesia | 24 hours postoperatively
  satisfaction from postoperative analgesia on a six-point Likert scale with 1 marked as minimal satisfaction and 6 as maximal satisfaction
first fluid intake | 24 hours postoperatively
  patients will be questioned regarding the time they had their first fluid intake
first solid intake | 24 hours postoperatively
  patients will be questioned regarding the time they had their first solid intake
hospitalization time | 96 hours postoperatively
  duration of hospital stay after surgery in hours
side effects intraoperatively | intraoperatively
  patients will be monitored for side-effects of the administered agents intraoperatively
side effects postoperatively | 48 hours postoperatively
  patients will be monitored for side-effects of the administered agents postoperatively

OTHER OUTCOMES:
time to emergence | up to 2-3 hours after start of surgery]
  time from sevoflurane discontinuation to first patient response (eye opening)
time to extubation | up to 2-3 hours after start of surgery]
  time from sevoflurane discontinuation to tracheal extubation

CONTACTS AND LOCATIONS:
Overall Officials: KASSIANI THEODORAKI, MD, PhD, DESA, Principal Investigator — Aretaieion University Hospital, National and Kapodistrian University of Athens, Greece
Locations (1):
- General Hospital of Athens, "Georgios Gennimatas", Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fletcher D, Martinez V. Opioid-induced hyperalgesia in patients after surgery: a systematic review and a meta-analysis. Br J Anaesth. 2014 Jun;112(6):991-1004. doi: 10.1093/bja/aeu137. PMID 24829420
- [Background] Forget P. Opioid-free anaesthesia. Why and how? A contextual analysis. Anaesth Crit Care Pain Med. 2019 Apr;38(2):169-172. doi: 10.1016/j.accpm.2018.05.002. Epub 2018 Sep 13. PMID 29775728
- [Background] Martin JL, Koodie L, Krishnan AG, Charboneau R, Barke RA, Roy S. Chronic morphine administration delays wound healing by inhibiting immune cell recruitment to the wound site. Am J Pathol. 2010 Feb;176(2):786-99. doi: 10.2353/ajpath.2010.090457. Epub 2009 Dec 30. PMID 20042674
- [Background] Ziemann-Gimmel P, Goldfarb AA, Koppman J, Marema RT. Opioid-free total intravenous anaesthesia reduces postoperative nausea and vomiting in bariatric surgery beyond triple prophylaxis. Br J Anaesth. 2014 May;112(5):906-11. doi: 10.1093/bja/aet551. Epub 2014 Feb 18. PMID 24554545
- [Background] Song JY, Choi H, Chae M, Ko J, Moon YE. The effect of opioid-free anesthesia on the quality of recovery after gynecological laparoscopy: study protocol for a prospective randomized controlled trial. Trials. 2021 Mar 12;22(1):207. doi: 10.1186/s13063-021-05166-z. PMID 33712080
- [Background] Ledowski T. Objective monitoring of nociception: a review of current commercial solutions. Br J Anaesth. 2019 Aug;123(2):e312-e321. doi: 10.1016/j.bja.2019.03.024. Epub 2019 Apr 30. PMID 31047645
- [Background] Frauenknecht J, Kirkham KR, Jacot-Guillarmod A, Albrecht E. Analgesic impact of intra-operative opioids vs. opioid-free anaesthesia: a systematic review and meta-analysis. Anaesthesia. 2019 May;74(5):651-662. doi: 10.1111/anae.14582. Epub 2019 Feb 25. PMID 30802933